CLINICAL TRIAL: NCT03957434
Title: Pilot Study Examining Feasibility and Effects of Physiotherapy Treatment Compared to Standard Usual Care in Gynecological Cancer Survivors With Urinary Incontinence
Brief Title: Physiotherapy Treatment for Gynecological Cancer Survivors With Urinary Incontinence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Institut Universitaire de Gériatrie de Montréal (Other); Jewish General Hospital (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and Associate Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-31-2017-1683
Record Dates: First submitted 2019-04-10; First posted 2019-05-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Cancer; Urinary Incontinence
Keywords: Pilot study; Gynecological cancer survivors; Urinary Incontinence; Physiotherapy
MeSH Terms: conditions — Urinary Incontinence | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Baseline evaluation - Randomization to physiotherapy or standard usual care (12 weeks) - Post-treatment evaluation
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiotherapy (Experimental): 12-weekly physiotherapy treatment sessions.
  Interventions: Other: Physiotherapy
- Standard usual care (No Intervention): Participants will be asked to continue the usual care established during the regular follow-up with their medical doctor for 12 weeks.

INTERVENTIONS:
Other: Physiotherapy — Education, pelvic floor muscle exercises with biofeedback and home exercises.
  Other Names: Pelvic floor rehabilitation
  Arms: Physiotherapy

SUMMARY:
The aims of this pilot study are to examine the feasibility and to explore the effects of a physiotherapy treatment compared to standard usual care in gynecological cancer survivors with urinary incontinence in preparation of a large randomized controlled study.

DETAILED DESCRIPTION:
Epidemiological studies demonstrated a growing number of gynecological cancer survivors, and this population is at great risk of developing pelvic floor dysfunction after cancer and its treatment. Representing the most prevalent pelvic floor dysfunction, urinary incontinence affects up to 70% of gynecological cancer survivors. International practice guidelines, in line with available meta-analysis, recommend physiotherapy as a first-line treatment to reduce urinary incontinence. However, there is limited evidence on its effectiveness in gynecological cancer survivors. Considering the current knowledge and the negative impacts of urinary incontinence, there is an urgent need to examine whether this population can benefit from this intervention in a pilot study, to conduct eventually a larger randomized controlled trial. The objectives of the present study are to examine the feasibility and to explore the effects of a physiotherapy treatment compared to standard usual care in gynecological cancer survivors with urinary incontinence. A total of 44 participants will be randomized to receive either physiotherapy or standard usual care (wait-list for physiotherapy). Baseline and post-treatment evaluations will be realized by a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* History of gynecological cancer (endometrial, cervical, vaginal or other parts of the uterus)
* Scheduled oncological treatments completed
* Stress or mixed urinary incontinence with a frequency of at least three urinary leakage per

Exclusion Criteria:

* Pelvic floor rehabilitation in the last year
* Other conditions interfering with assessment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2025-10-16 (Estimated); Study Completion 2025-10-16 (Estimated)

PRIMARY OUTCOMES:
Adherence rates | Baseline to 2-week post-treatment evaluation
  To determine acceptability by assessing adherence to exercises.
Retention rate | Baseline to 2-week post-treatment evaluation
  To determine feasibility by evaluating attrition.

SECONDARY OUTCOMES:
Change from baseline in number of urinary leaks | Baseline to 2-week post-treatment
  7-day voiding schedule will be used to evaluate the reduction of urinary leakage.
Change from baseline in symptoms of pelvic floor dysfunction | Baseline to 2-week post-treatment evaluation
  To explore changes in pelvic floor symptoms (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form ranging from 0 to 21), a high score represents high pelvic floor symptoms.
Change from baseline in pelvic floor muscle function | Baseline to 2-week post-treatment evaluation
  To explore changes in pelvic floor muscle function at rest and during contraction (dynamometry).
Change from baseline in pelvic floor muscle morphometry | Baseline to 2-week post-treatment evaluation
  To explore changes in pelvic floor muscle function at rest and during contraction (ultrasound).
Change from baseline in sexual function | Baseline to 2-week post-treatment evaluation
  To explore changes in sexual function (Female Sexual Function Index ranging from 2 to 36), a low score represents a low sexual function.
Change from baseline in quality of life | Baseline to 2-week post-treatment evaluation
  To explore changes in quality of life (European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire ranging from 0 to 100), a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / quality of life represents a high quality of life and a high score for a symptom scale / item represents a high level of symptomatology / problems.
Patient's global impression of change | Baseline to 2-week post-treatment evaluation
  To determine patient self-reported improvement (Patient's Global Impression of Change ranging from "very much worse" to "very much improved" on a 7-point scale.
Rate of adverse events | Baseline to 2-week post-treatment evaluation
  To document any adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche du Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada